CLINICAL TRIAL: NCT01379573
Title: Preventive Approach to Congenital Heart Block With Hydroxychloroquine
Acronym: PATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-00369
Record Dates: First submitted 2011-06-16; First posted 2011-06-23 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Congenital Heart Block; Neonatal Lupus; Autoantibody-Associated Heart Block
Keywords: hydroxychloroquine; Plaquenil; congenital heart block; neonatal lupus; systemic lupus erythematosus; Sjogren's syndrome; autoantibodies; SSA/Ro; SSB/La; autoimmunity; pregnancy; immunoglobulin
MeSH Terms: conditions — Congenital heart block; Neonatal Systemic lupus erythematosus; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Autoimmune Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pregnant women with previous child with cardiac neonatal lupus (Experimental): 400 mg/day Hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Nineteen women meeting eligibility criteria will receive 400mg per day of HCQ beginning as soon as pregnancy is established and informed consent obtained. Mothers already on HCQ will remain on 400mg, or escalate to 400mg if on 200mg. Hydroxychloroquine is taken in 200mg pill form - 400mg = 2 200mg pills.
  Other Names: Plaquenil

SUMMARY:
Women with antibodies to proteins called SSA/Ro and or SSB/La face a 2% chance of having a child with a life threatening heart condition regardless of whether they have very active lupus, are in remission, or have only vague symptoms. This heart problem is referred to as congenital heart block (the most serious being third degree complete block) and represents damage thought to be caused by these autoantibodies. The heart beats abnormally slowly and almost all children require permanent pacemakers before the age of 20. Importantly, women who have had one child with heart block have a ten-fold higher risk of having another child with the same heart condition. Unfortunately, even close monitoring by special techniques during pregnancy does not reverse complete heart block once it is observed. Thus, treatments aimed at prevention are critical. This study will evaluate for the first time whether hydroxychloroquine, a drug used by many patients with SLE, prevents the development of this heart condition. Data from laboratory experiments suggests that this drug, which crosses the placenta, may decrease the inflammation initiated by the passage of anti-Ro antibodies to the fetus. The study uses a Simon's 2-Stage design, and plans to enroll 19 patients in Stage 1 and 35 patients in Stage 2 if Stage 1 is successful. Patients can already be on hydroxychloroquine or will be started as soon as pregnancy is confirmed. The hope is that fewer than 3 cases of heart block will occur in Stage 1, and fewer than 6 cases will occur out of all 54 patients if Stage 2 is reached. The results of this study are expected to become an integral part of the counseling of women with anti-Ro/La antibodies who are considering pregnancy.

DETAILED DESCRIPTION:
One of the strongest clinical associations with autoantibodies directed to components of the Ro/La ribonucleoprotein complex is the development of congenital heart block (CHB) in an offspring, an alarming prospect facing 2% of primigravid mothers with these reactivities. The risk is 10-fold higher in women who have had a previously affected child. Despite the attempt of large multicenter studies to forestall disease by serial in utero monitoring, irreversible block and extensive myocardial injury have been documented within 7 days of a normal rhythm and PR interval. CHB is associated with a substantial mortality and morbidity. Two recent prospective studies (20 mothers from U.S. and 15 from Europe) utilizing an identical protocol of IVIG at replacement doses demonstrated 1) this intervention does not prevent the recurrence of CHB 2) the recurrence rate of 17-18% is robust 3) recruitment of patients is feasible. During the time period of the IVIG trials, basic science exploring the pathogenesis of disease supported the notion that Toll Like Receptor (TLR) signaling following ligation of ssRNA (hY3) complexed to the Ro protein contributes to fibrosis. This observation led to in vitro studies addressing inhibition of endosomal acidification by chloroquine and subsequent translation to patients by evaluating the use of hydroxychloroquine (HCQ) in an extensive retrospective chart review. The combined data suggest efficacy of HCQ. Accordingly, the goal of this study is to: To determine whether hydroxychloroquine use during pregnancy prevents CHB in a high risk population. The trial is open-label and employs the Simon's 2-stage optimal design to allow for early stopping due to absence of treatment efficacy. The first stage requires 19 subjects. Despite the rarity of disease and the requirement of a previous CHB child, based on the US Research Registry for Neonatal Lupus, this proposal is feasible. If 3 or more mothers have a child with 2nd or 3rd degree CHB, the study is terminated after the first stage. If this does not occur, funds will be sought to enroll an additional 35 mothers in the second stage for a total of 54 subjects. Treatment will be considered efficacious if fewer than 6 mothers of 54 have a child with advanced CHB. With this design, the study has 90% power to conclude that hydroxychloroquine is preventive if the true recurrence rate with the treatment is 5%. In addition, the probability of rejecting the treatment for further study is 95% if the true recurrence rate is 18%. Serial echocardiograms (monitor PR interval) and blood drawing (IFNƒÑƒnsignatures, antibody titers) will be included in the protocol. The results of this study are expected to become an integral part of the counseling of women with anti-SSA/Ro-SSB/La antibodies who are considering pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers must have anti-Ro and/or anti-La Ab documented in the NYU immunology laboratory (CLIA-approved), which utilizes an ELISA as well as reactivity on ELISA to at least one of three recombinant antigens (48La, 52Ro, 60Ro, JB laboratory).
2. Mothers must have a previous child with cardiac NL, defined herein as: the presence of heart block (1st, 2nd, or 3rd degree) documented by electrocardiogram (EKG), echocardiogram, pacemaker, or statement in the medical record, and/or; presence of cardiac injury, which specifically includes autopsy evidence of a mononuclear infiltrate in the endocardium, myocardium, and pericardium and/or EFE on echocardiogram always associated with cardiac dysfunction. In PITCH, we included women with a prior child with rash; however, recent data generated from the RRNL suggest that recurrence of CHB following rash is 11%, not 18% [34]. Thus, inclusion of previous rash could lead to a falsely lowered recurrence rate, and will therefore be excluded.
3. Intrauterine pregnancy ≤10 weeks.
4. Mother may be taking ≤20 mg prednisone because, in our experience, CHB has developed in the presence of this dose.
5. Mother may be asymptomatic, or have a rheumatic disease such as SLE or SS. Maternal health status has not been considered an influence on the development of CHB.
6. Mother may or may not already be taking HCQ. This latter point was discussed with Dr. Nathalie Costedoat-Chalumeau, who has published extensively on measurement of HCQ. While it might be optimal for the mothers anticipating enrollment in the study to all have been on HCQ prior to conception, this is impractical. Some may never achieve pregnancy and not want to take HCQ unless they conceive (especially those asymptomatic). On the other hand, women with SLE are likely to already be on HCQ and it would limit enrollment to exclude these patients if all must initiate HCQ only at enrollment in the first trimester. Although the accepted dogma is that HCQ requires several months for maximal efficacy in treating rheumatic disease, it is unknown whether this would apply to transplacental passage or fetal levels (which are impossible to measure). Dr. Costedoat-Chalumeau suggests that HCQ is probably a three compartment model which includes the circulation, tissues and cells. In the circulation, the half life is approximately 7 days and in the tissues, it is 40 days. In Dr. Costedoat-Chalumeau's experience, steady state blood levels of HCQ are achieved in 4-6 weeks. Thus, dosing the mother no later than 10 weeks gestation should provide sufficient fetal exposure before the vulnerable period of CHB which is generally accepted to span 18-24 wks. Furthermore, the placenta has to be formed for HCQ to gain access to the fetus and it may be effective quickly for the biology we are considering.

Exclusion Criteria:

1. Mother does not have Ab to Ro or La.
2. Identification of any of the following structural lesions considered causal for CHB, i.e., those that could account for block because of fibrous disruption between the atrium and AV node or due to absence of the penetrating bundles of the AV node:

   * atrioventricular septal defects;
   * b) single ventricle
   * c) developmental tricuspid valve disease;
   * d) L-transposition of the great arteries;
   * e) heterotaxia.
3. Mother is taking any glucocorticoids. Although unlikely to be preventative, the use of steroids may confound the interpretation of results. The final point of intense discussion centered around whether another exclusion should be the use of HCQ in the first pregnancy in which CHB occurred. While one could argue that in these mothers HCQ was not effective and perhaps will not be again, this assumption remains speculative and thus prior absence of efficacy of HCQ will not constitute an exclusion criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill P Buyon, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Friedman DM, Kim M, Costedoat-Chalumeau N, Clancy R, Copel J, Phoon CK, Cuneo BF, Cohen R, Masson M, Wainwright BJ, Zahr N, Saxena A, Izmirly PM, Buyon JP. Electrocardiographic QT Intervals in Infants Exposed to Hydroxychloroquine Throughout Gestation. Circ Arrhythm Electrophysiol. 2020 Oct;13(10):e008686. doi: 10.1161/CIRCEP.120.008686. Epub 2020 Sep 9. PMID 32907357
- [Derived] Izmirly P, Kim M, Friedman DM, Costedoat-Chalumeau N, Clancy R, Copel JA, Phoon CKL, Cuneo BF, Cohen RE, Robins K, Masson M, Wainwright BJ, Zahr N, Saxena A, Buyon JP. Hydroxychloroquine to Prevent Recurrent Congenital Heart Block in Fetuses of Anti-SSA/Ro-Positive Mothers. J Am Coll Cardiol. 2020 Jul 21;76(3):292-302. doi: 10.1016/j.jacc.2020.05.045. PMID 32674792

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women With Previous Child With Cardiac Neonatal Lupus: 400 mg/day Hydroxychloroquine
  Hydroxychloroquine: women meeting eligibility criteria will receive 400mg per day of HCQ beginning as soon as pregnancy is established and informed consent obtained. Mothers already on HCQ will remain on 400mg, or escalate to 400mg if on 200mg. Hydroxychloroquine is taken in 200mg pill form - 400mg = 2 200mg pills.
Period: Overall Study
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Started | 74
Completed | 63
Not Completed | 11
Not completed — Lost to Follow-up | 1
Not completed — Screen Failure | 10

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Age, Continuous [Mean (Full Range); unit: years] | 32.7 [28.8 to 36.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 45
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 62
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Advanced Heart Block
Description: Echocardiogram reveals 2nd or 3rd degree AV block
Time Frame: After enrollment at 16-18 weeks gestation, then weekly until 26 weeks, biweekly to 34 weeks, at birth (approximately 9 months), and at one year follow up (approximately 21 months from enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 5

2. Secondary Outcome: Prolonged PR Interval (>150msec)
Description: EKG at birth must confirm 1st degree AV block. It is also possible that a fetus developing 1st degree block on study medication might have developed more advanced block in the absence of study medication.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 0

3. Secondary Outcome: Any Sign of Myocardial Injury, Without Change in Cardiac Rate or Rhythm
Description: a) shortening fraction <28% = 2 SD below normal mean or qualitatively reduced systolic function; b) cardio-thoracic ratio >0.33; c) hydropic changes; d) moderate/severe tricuspid regurgitation.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 0

4. Secondary Outcome: Echocardiographic Densities Consistent With EFE Confirmed Postnatally
Description: (see title)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 0

5. Secondary Outcome: Fetal Death Not Related to Cardiac Dysfunction
Description: An autopsy with full evaluation of the heart will be encouraged but cannot be mandated. If AV block or evidence of a cardiomyopathy can be "proven," then these will provide the basis for final categorization. If not possible, the death will not be considered a recurrence rate but will be reported.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 0

6. Secondary Outcome: Cutaneous Neonatal Lupus
Time Frame: Up to 15 months (at birth - 9 months, and 6 months thereafter)
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 4

7. Secondary Outcome: Prematurity
Description: (gestational age <37 weeks at birth)
Time Frame: At birth (approximately 9 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 9

8. Secondary Outcome: Birth Weight <10% in the Context of Gestational Age
Time Frame: At birth (approximately 9 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 1

9. Secondary Outcome: Abnormal Fluid Collection
Time Frame: At birth (approximately 9 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
Number analyzed (Participants) | 63
Participants | 0

ADVERSE EVENTS:
Time Frame: From time of enrollment to six months after delivery.
Arm/Group | Pregnant Women With Previous Child With Cardiac Neonatal Lupus
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 11/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnant Women With Previous Child With Cardiac Neonatal Lupus (N=63)
Maternal rash (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Spontaneous miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Severe itching (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Fall (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Placental abruption (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Placenta previa (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abnormal neonatal liver function test lab values (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Right bundle branch block (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT01379573/Prot_SAP_000.pdf